CLINICAL TRIAL: NCT02827539
Title: A Prospective, Randomized Study of LessRay Enhanced Versus Standard Fluoroscopic Visualization in Surgical Placement of Spinal Cord Stimulator Epidural Array
Brief Title: A Prospective Study of LessRay Enhanced Versus Standard Fluoroscopic Visualization in Surgical Placement of Spinal Cord Stimulator
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in resources to support study activities
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Pro00070805
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Fluoroscopy for Spine Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Research (Other): If the patient is randomized to the Research Arm, the physician will begin the procedure utilizing LessRay enhanced fluoroscopic images.
  Interventions: Device: LessRay
- Control (Other): For patients in the control arm standard fluoroscopy will be used with the C-arm set to the conventional full dose setting
  Interventions: Device: Standard Fluoroscopy

INTERVENTIONS:
Device: LessRay — A software device has been developed that combines the benefits of reduced radiation associated with low-dose and/or pulse settings while preserving and possibly offering enhanced resolution. LessRay is a software device that is viewed on a separate monitor next to the fluro screen of the C-arm.
  Arms: Research
Device: Standard Fluoroscopy — For control arm, patients will receive the standard fluoroscopy for imaging.
  Arms: Control

SUMMARY:
The purpose of this study is to gather information comparing LessRay Enhanced fluoroscopy with the current standard of fluoroscopy. This research is being conducted to demonstrate the utility and effectiveness of LessRay Enhanced fluoroscopy during surgical placement of a spinal cord stimulator epidural array.

DETAILED DESCRIPTION:
The purpose of this prospective, randomized single center study is to assess the ability of LessRay to decrease overall radiation exposure during surgical placement of a spinal stimulator. A secondary objective is to analyze the efficacy of utilizing enhanced low radiation imaging in a fluoroscopically intensive pain procedure.

The population group will be 65 patients from Duke University Medical Center and Duke Raleigh Hospital who meet the medical criteria for the surgical placement of a spinal cord stimulator epidural array. They will be divided equally into 2 arms: Research and Control and randomized by a non-surgeon on the study team. That information will be recorded and placed in a sealed envelope. On the day of surgery the envelope will be delivered to the OR and opened following "time-out". At the time the envelope is opened in the OR the patient is acknowledged to be evaluable for failure or success of LessRay during the surgical procedure if they are in the research arm. The control arm cohort will proceed with the surgery as typical without LessRay.

The data from the two groups (Research vs. Control) will be analyzed using a two tailed t-test with p<.05. The risks associated specifically with the implementation of this study are with respect to loss of confidentiality. Every effort will be made to keep the information confidential

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults of any ethnicity
* At least 18 years-old but without an upper age limit
* Subject is willing to provide informed, written consent to participate in this study
* Subject meets the medical criteria for surgical placement of a spinal cord stimulator epidural array (e.g. not pregnant)

Exclusion Criteria:

* Less than 18 years of age. For both physicians involved in the study, standard of care Spinal Cord Stimulator placement is not done for those patients under 18 years of age as the literature does not show that the procedure helps in back pain of this cohort of patients
* Unable to provide informed, written consent
* Pregnant women as pregnancy makes them ineligible to undergo a surgical placement of a spinal cord stimulator
* Prior placement of a spinal cord stimulator epidural array or previous thoracic spine surgery, which could potentially make placement more difficult
* Enrollment in another study, which would prohibit participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

PRIMARY OUTCOMES:
Radiation exposure | During the surgery
  Radiation dose provided to the patient in each arm of the study will be recorded
Efficacy as measured by image resolution | During the surgery
  Image resolution provided by the radiation dose used in each arm of the study will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nandan Lad, MD, PhD, Principal Investigator — Duke UMC
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: 1. Food and Drug Administration. 2010. "White Paper: Initiative to Reduce Unnecessary Radiation Exposure from Medical Imaging." — http://www.fda.gov/Radiation-EmittingProducts/RadiationSafety/RadiationDoseReduction/ucm199994.htm